CLINICAL TRIAL: NCT02213887
Title: A Pilot Study to Determine if Pantoprazole Modifies Steady-State Plasma Concentrations of Orally Administered Psychotropic Medications
Brief Title: Study of the Effects of Pantoprazole on Levels of Prescribed Psychiatric Medications
Acronym: PK-PPI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ric Procyshyn, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H14-01095
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Psychotic Disorders; Gastroesophageal Reflux
Keywords: Drug Interactions; Pantoprazole; Proton Pump Inhibitors; Psychotropic Drugs; Antipsychotic Agents; Aripiprazole; Asenapine; Clozapine; Lurasidone; Olanzapine; 9-hydroxy-risperidone; Quetiapine; Risperidone; Ziprasidone; Valproic Acid; Lithium; Gastrins; Psychotic Disorders; Gastroesophageal Reflux
MeSH Terms: conditions — Psychotic Disorders; Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Start Pantoprazole (Experimental): Participants have been diagnosed with gastroesophageal reflux disease but have not started pharmacological treatment.
  Intervention: Days 2-8
  Interventions: Drug: Pantoprazole
- Stop Pantoprazole (Experimental): Participants have been taking pantoprazole for more than 8 weeks and are asymptomatic for gastroesophageal reflux disease.
  Intervention: Days 2-8
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — 40 mg PO QAM
  Other Names: Pantoloc; Protonix
  Arms: Start Pantoprazole
Drug: Pantoprazole — 0 mg PO QAM
  Other Names: Pantoloc; Protonix
  Arms: Stop Pantoprazole

SUMMARY:
The purpose of this 9-day study is to determine if:

1. Pantoprazole modifies the steady-state plasma concentrations of orally administered psychotropic medications including valproic acid, lithium, and second-generation antipsychotics (i.e., aripiprazole, asenapine, clozapine, lurasidone, olanzapine, paliperidone, quetiapine, risperidone, ziprasidone)
2. Serum gastrin levels change within a week of starting or stopping pantoprazole

DETAILED DESCRIPTION:
Individuals with psychiatric diagnoses may be predisposed to gastroesophageal reflux disease because of the widespread use of alcohol, cigarettes, and certain psychotropic drugs in this population. Consequently, they are often prescribed proton pump inhibitors. To our knowledge, no studies have been conducted to determine the effects of proton pump inhibitors on plasma levels of psychotropic drugs. The present clinical study will assess the effects of pantoprazole on the pharmacokinetics of valproic acid, lithium, and second-generation antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be fluent in English
* Participants with a psychiatric diagnosis and currently treated with one or more of the following medications: valproic acid, lithium, or a second-generation antipsychotic (i.e., aripiprazole, asenapine, clozapine, lurasidone, olanzapine, paliperidone, quetiapine, risperidone, or ziprasidone)
* Participants on a stable dose of valproic acid, lithium, and/or a second-generation antipsychotic for a sufficient period of time that ensures they are at steady state
* Participants with symptoms of gastroesophageal reflux disease (GERD) that would benefit from treatment with pantoprazole or participants currently treated for GERD with pantoprazole for more than 8 weeks and are currently symptom free.

Exclusion Criteria:

* Participants that are hypersensitive to pantoprazole
* Pregnant or lactating women
* Women of childbearing age not using reliable contraception
* Any postsurgical complications of the gastrointestinal tract that might impair absorption
* Clinically relevant abnormalities of laboratory parameters
* Participants treated with another acid suppressing agent (e.g., H2 receptor antagonists, antacids, alginates, etc)
* Participants treated with atazanavir, delavirdine, erlotinib, nelfinavir, and/or posaconazole

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in steady-state plasma concentrations of psychotropic medication(s) at Days 2, 5, and 9. | Days 1(baseline), 2 , 5, and 9
  Pharmacokinetic outcome measures often require multiple measurement over time. On Day 1, baseline steady-state plasma concentration of psychotropic medication(s) will be determined. On Days 2, 5, and 9, steady-state plasma concentration of psychotropic medication(s) will be determined and compared to baseline

SECONDARY OUTCOMES:
Change from baseline in fasting serum gastrin concentrations at Day 9. | Days 1 (baseline) and 9
  On Day 1, baseline fasting serum gastrin concentration will be determined. On Day 9, fasting serum gastrin concentration will be determined and compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ric M. Procyshyn, Ph.D, Principal Investigator — University of British Columbia; Alasdair Barr, Ph.D, Study Director — University of British Columbia; William Honer, MD, Study Director — University of British Columbia; Randall White, MD, Study Director — University of British Columbia
Locations (1):
- UBC Hospital - Detwiller Pavilion, Vancouver, British Columbia, Canada